CLINICAL TRIAL: NCT02360319
Title: A Cluster Randomized, Multi-center, Parallel-group, Rater-blind Study Comparing Treatment With Aripiprazole Once Monthly and Treatment as Usual on Effectiveness in First Episode and Early Phase Illness in Schizophrenia
Brief Title: Comparison of a Long-acting Injectable Antipsychotic vs Clinician's Choice Early in Treatment to Break the Cycle of Relapse in Early Phase Schizophrenics
Acronym: PRELAPSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanguard Research Group (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: COL.AOM.2013.005
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia
Keywords: First episode or recent onset
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinician's Choice (Active Comparator): Prescribers are not limited in the choice of treatment they can administer to their clients to alleviate the symptoms of schizophrenia. Any FDA approved antipsychotic agent can be used. Clients in the study wil be followed for 2 years
  Interventions: Drug: Any FDA approved antipsychotic agent
- Aripiprazole Once Monthly (Experimental): Aripiprazole long acting injectable formulation, 400mg per dose is to be administered once monthly. Clients in the study will be followed for 2 years
  Interventions: Drug: aripiprazole long acting injectable formulation

INTERVENTIONS:
Drug: Any FDA approved antipsychotic agent — Investigators are free to choose the most appropriate treatment for their clients
  Arms: Clinician's Choice
Drug: aripiprazole long acting injectable formulation
  Arms: Aripiprazole Once Monthly

SUMMARY:
The goal of this project is to show that the best possible option for preventing relapses in patients suffering from first episode (<1 year of anti-psychotic medication) or early phase (< 5 years of lifetime exposure to anti-psychotic medication) schizophrenia is by enhancing medication adherence. The study is designed to answer the question of whether the use of long-acting injectable (LAI) antipsychotics early in the course of treatment can break the cycle of frequent relapse that affects so many patients with early phase schizophrenia. The participating research sites (not individual patients) will be randomly assigned to either medication prescribed by their treating physician (with no restrictions) or to a regimen that involves a monthly long acting injectable antipsychotic. The sites will be assigned on a one to one basis to either of the arms taking into account types of patient population and geographical area. Patients enrolled in the study will participate in regular assessments either over the phone or in person and be followed for a period of 2 years. The primary outcome measure is time to first hospitalization.

DETAILED DESCRIPTION:
Approximately 40 U.S. sites will participate in the study in order to enroll approximately 500 patients over a year period. They will be recruited into two cohorts - the first episode cohort and the early phase (EP) cohort, with approximately 250 patients in each cohort. Enrollment of patients will be discontinued when the appropriate number for the target for each cohort is reached.

After providing written informed consent, patients will be screened for general eligibility by the clinical team at the site. Basic demographic data will be collected to determine suitability for inclusion into the study. The site will complete an information interview comprising data regarding symptomology and history, but the diagnosis of schizophrenia will fall to a centralized, remote blinded rater to enable consistency for eligibility.

Prescribers at sites in the clinician's choice arm can treat the patients in the manner most appropriate for that individual. Prescribers at sites in the Aripiprazole Once Monthly arm monthly will prescribe and administer the medication according to recommendations contained in the product labeling.

For a period of 2 years all subjects will receive bimonthly calls inquiring about visits to emergency rooms and hospitalization. At 4 month intervals information on use of services, insurance status, work, school attendance, and other service use outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Are able to provide written informed consent Have a confirmed diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual (DSM) 5 criteria using the SCID (Structured Clinical Interview for DSM disorders) Are between the ages of 18 and 35, inclusive Have the following history with antipsychotic medications

1. First episode subjects: < 1 year of lifetime exposure to antipsychotic medication and only one episode of psychosis
2. EP subjects: between 1 year and 5 years of lifetime exposure to antipsychotic medication or subjects with < 1 year of lifetime antipsychotic medication and more than one episode of psychosis.

For LAI subjects: Must be willing to accept an injectable form of treatment

Exclusion Criteria:

Have a current primary DSM-5 diagnosis other than schizophrenia, including schizophreniform disorder, schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, and amnestic or other cognitive disorders.

For LAI sites only - have a known allergy or intolerance to aripiprazole, or a past negative response to aripiprazole that is not explained by nonadherence Be pregnant or lactating Have any unstable medical condition that, in the opinion of the investigator, would be detrimental to the subject or would confound the results of the study Subjects in the MRI subset only- presence of any metal implants, pacemakers, irremovable prosthetic devices, or other devices or situations that may preclude imaging

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 489 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Kane, M.D., Principal Investigator — Northwell Health
Locations (39):
- United States (39):
  - La Frontera, Tucson, Arizona
  - San Fernando Mental Health Center, Granada Hills, California
  - Stanford School of Medicine, Palo Alto, California
  - Henderson Behavioral Health, Fort Lauderdale, Florida
  - Meridian Behavioral Healthcare, Gainesville, Florida
  - U. of Florida College of Medicine, Jacksonville, Florida
  - LifeStream Behavioral Center, Leesburg, Florida
  - Suncoast Center, St. Petersburg, Florida
  - Apalachee Center, Inc., Tallahassee, Florida
  - Jerome Golden Center for Behavioral Health, West Palm Beach, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Chestnut Health Systems, Granite City, Illinois
  - University of Iowa Psychiatry Research, Iowa City, Iowa
  - Corrigan Mental Health Center, Fall River, Massachusetts
  - U. Mass Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Early Treatment and Cognitive Health, East Lansing, Michigan
  - Cherry Street Health Services, Grand Rapids, Michigan
  - WMU School of Medicine, Kalamazoo, Michigan
  - Community Mental Health for Central Michigan, Mount Pleasant, Michigan
  - Muskegon County Community Mental Health, Muskegon, Michigan
  - Saint Louis University CRU, St Louis, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - The Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Healthy Perspectives, Nashua, New Hampshire
  - New Bridge Medical Center, Paramus, New Jersey
  - Carolina Behavioral Care, Durham, North Carolina
  - Central Community Health Board of Hamilton Co., Cincinnati, Ohio
  - The Counseling Center of Wayne and Holmes Counties, Wooster, Ohio
  - PeaceHealth Medical Group, Eugene, Oregon
  - Carey Counseling Center, Huntingdon, Tennessee
  - Spindletop Center, Beaumont, Texas
  - Baylor College of Medicine, Houston, Texas
  - MHC Community Healthcore, Longview, Texas
  - The Center for Health Care Services, San Antonio, Texas
  - Psychiatric & Behavioral Solutions, Salt Lake City, Utah

REFERENCES:
- [Derived] Kane JM, Schooler NR, Marcy P, Correll CU, Achtyes ED, Gibbons RD, Robinson DG. Effect of Long-Acting Injectable Antipsychotics vs Usual Care on Time to First Hospitalization in Early-Phase Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Dec 1;77(12):1217-1224. doi: 10.1001/jamapsychiatry.2020.2076. PMID 32667636
- [Derived] Kane JM, Schooler NR, Marcy P, Achtyes ED, Correll CU, Robinson DG. Patients With Early-Phase Schizophrenia Will Accept Treatment With Sustained-Release Medication (Long-Acting Injectable Antipsychotics): Results From the Recruitment Phase of the PRELAPSE Trial. J Clin Psychiatry. 2019 Apr 23;80(3):18m12546. doi: 10.4088/JCP.18m12546. PMID 31050233

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole Once Monthly: Aripiprazole long acting injectable formulation, 400mg per dose is to be administered once monthly. Clients in the study will be followed for 2 years
  aripiprazole long acting injectable formulation
Period: Overall Study
Arm/Group | Clinician's Choice | Aripiprazole Once Monthly
Started | 255 | 234
Completed | 167 | 173
Not Completed | 88 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician's Choice | Aripiprazole Once Monthly | Total
Number analyzed (Participants) | 255 | 234 | 489
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (4.1) | 25.7 (4.3) | 25.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 62 | 121
  Male | 196 | 172 | 368
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 104 | 109 | 213
  White | 91 | 80 | 171
  More than one race | 45 | 39 | 84
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 255 | 234 | 489

OUTCOME MEASURES:

1. Primary Outcome: Time to First Hospitalization
Description: Assessments are done using best available data and patient interviews
Time Frame: Hospitalizations assessed every 2 months from baseline to Month 24
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Clinician's Choice | Aripiprazole Once Monthly
Number analyzed (Participants) | 255 | 234
days | 530.6 [497.3 to 563.9] | 613.7 [582.3 to 645.1]

2. Secondary Outcome: Total Number of Psychiatric Hospitalizations Per Treatment Arm
Description: Assessments are completed using best available data and patient interviews
Time Frame: Measured every 2 months from baseline to month 24
Population: Intent to treat
Measure: Number; unit: Hospitalizations
Arm/Group | Clinician's Choice | Aripiprazole Once Monthly
Number analyzed (Participants) | 255 | 234
Hospitalizations | 208 | 133

3. Secondary Outcome: Brief Psychotic Rating Scale (BPRS) Total Score
Description: The Brief Psychotic Rating Scale is an 18 item scale where each item is rated 1-7, the minimum total score is 18 and the maximum total score is 126. Higher scores indicate more severe symptoms.
Time Frame: Measured at Month 12 and Month 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Clinician's Choice | Aripiprazole Once Monthly
Number analyzed (Participants) | 255 | 234
Scores on a scale
  Baseline | 35.59 (9.40) | 35.45 (9.27)
  Month 12 | 30.7 (8.73) | 31.31 (9.32)
  Month 24 | 30.73 (8.86) | 30.87 (9.13)

4. Secondary Outcome: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Sum of Scores
Description: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a 12 item scale with a total score range of 0 to 321 with higher scores indicating better cognitive functioning
Time Frame: Measured at Month 12 and Month 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Clinician's Choice | Aripiprazole Once Monthly
Number analyzed (Participants) | 255 | 234
Scores on a scale
  Baseline | 182.4 (33.1) | 177.7 (35.4)
  Month 12 | 189.2 (34.9) | 178.2 (34.9)
  Month 24 | 194.1 (33.2) | 180.8 (33.6)

5. Secondary Outcome: Quality of Life (QLS) Total Score
Description: Quality of Life (QLS) is a 21 item scale where each item is rated from 0 to 7, the minimum score is 0 and the maximum score is 126 with higher scores indicating better overall functioning.
Time Frame: Measured at Month 12 and Month 24
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Clinician's Choice | Aripiprazole Once Monthly
Number analyzed (Participants) | 255 | 234
Scores on a scale
  Baseline | 63.60 (19.36) | 58.40 (19.83)
  Month 12 | 68.45 (23.13) | 65.02 (21.60)
  Month 24 | 62.21 (24.54) | 70.05 (24.28)

ADVERSE EVENTS:
Time Frame: All Adverse Events, regardless of relationship to study drug or procedure, were collected beginning from the time the subject signs the study Informed Consent Form through the last Visit, scheduled at 104 weeks following the Baseline Visit. Serious AEs were collected for 30 days after the last dose or at the Follow-up Visit, whichever comes later.
Arm/Group | Clinician's Choice | Aripiprazole Once Monthly
All-Cause Mortality (participants affected / at risk) | 2/255 | 0/234
Serious Adverse Events (participants affected / at risk) | 104/255 | 68/234
Other Adverse Events (participants affected / at risk) | 161/241 | 169/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinician's Choice (N=255) | Aripiprazole Once Monthly (N=234)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Psychiatric hospitalization/illness (Psychiatric disorders) | 96 (231) | 60 (143) — Worsening of psychosis or other psychiatric condition
Jail (Social circumstances) | 2 (2) | 0 (0)
Serious psychiatric event not requiring hospitalization (Psychiatric disorders) | 2 (2) | 3 (3)
Confusion (General disorders) | 1 (1) | 0 (0)
Cholecystectomy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abcess (Infections and infestations) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Angina (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 2 (5)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lactation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Drug Overdose (Social circumstances) | 0 (0) | 1 (1)
Chest laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinician's Choice (N=241) | Aripiprazole Once Monthly (N=222)
Weight Gain (Metabolism and nutrition disorders) | 47 (47) | 32 (32)
Depression (Psychiatric disorders) | 20 (20) | 23 (23)
Anxiety (Psychiatric disorders) | 15 (15) | 27 (27)
Hyperprolactemia (Endocrine disorders) | 31 (31) | 9 (9)
Elevated cholesterol levels (Cardiac disorders) | 24 (24) | 15 (15)
Hepatic enzyme abnormalities (Hepatobiliary disorders) | 22 (22) | 15 (15)
Insomnia (Psychiatric disorders) | 17 (17) | 19 (19)
Hypertension (Cardiac disorders) | 18 (18) | 12 (12)
Somnolence (Psychiatric disorders) | 11 (11) | 16 (16)
Hostility/aggression (Psychiatric disorders) | 7 (7) | 16 (16)
Tachycardia (Cardiac disorders) | 12 (12) | 7 (7)
Restlessness (Nervous system disorders) | 2 (2) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT02360319/Prot_SAP_000.pdf